CLINICAL TRIAL: NCT00384735
Title: An Adequate Cost Effective Follow Up Protocol For Bone & Soft Tissue Sarcomas - A Prospective Randomized Trial
Acronym: TOSS
Status: Completed | Type: Observational
Sponsor: Terry Fox Foundation (Other)
Collaborators: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Ajay Puri, Professor, Terry Fox Foundation
Other Study IDs: TOSS
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Sarcoma
Keywords: bone tumor; soft tissue tumor
MeSH Terms: conditions — Sarcoma; Bone Neoplasms; Soft Tissue Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1A: Intensive - 3 monthly follow up
- 1B: Intensive - 6 monthly follow up
- IIA: Cost Effective - 3 monthly follow up
- IIB: Cost Effective - 6 monthly follow up

SUMMARY:
The purpose of this study is to evaluate the impact on overall survival of an intensive follow-up protocol (as practiced today at TMH) against a more cost effective follow-up protocol in patients operated for extremity sarcoma.

DETAILED DESCRIPTION:
Follow up studies are performed for a variety of reasons. The detection of a recurrence of the index lesion is the foundation of surveillance. Detection of other medical conditions is a secondary benefit. Psychologically, follow up testing can serve as a source of reassurance. Whether an increased frequency of follow up and the use of various expensive imaging modalities for screening and early detection of recurrence actually results in improving overall survival of patients with extremity sarcomas is a question that remains as yet unanswered. Currently followed post -operative surveillance regimes are empirical and vary widely from centre to centre. Allocation of limited health funding should be guided by evidence based recommendations rather than empirical beliefs. An ideal surveillance regime should meet the criteria of easy implementation, accuracy and cost effectiveness.

In a vast country like India where patients often travel thousands of kilometers in their search for quality medical care the frequency of routine follow up visits is as important as studying the role of expensive screening modalities while drawing up guidelines for cost effective follow up strategies.

This study, a prospective randomized controlled trial, attempts to outline guidelines regarding the role of follow up vis a vis frequency and the use of various imaging modalities for early detection of recurrence in improving overall survival of patients with extremity sarcomas.

ELIGIBILITY:
Inclusion Criteria:

1. Patients operated for primary or recurrent extremity bone & soft tissue sarcomas.(both limb salvage and amputations)
2. Non Metastatic at presentation.
3. Patients reliable for follow-up.

Exclusion Criteria:

1. Non-extremity sarcomas.
2. Metastatic at presentation
3. Patients unreliable for follow up.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients operated for primary or recurrent extremity bone & soft tissue sarcomas
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2010-06-30 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Minimum 2 years

SECONDARY OUTCOMES:
Disease free survival | Minimum 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ajay Puri, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

REFERENCES:
- [Derived] Puri A, Gulia A, Hawaldar R, Ranganathan P, Badwe RA. Does intensity of surveillance affect survival after surgery for sarcomas? Results of a randomized noninferiority trial. Clin Orthop Relat Res. 2014 May;472(5):1568-75. doi: 10.1007/s11999-013-3385-9. Epub 2013 Nov 19. PMID 24249538